CLINICAL TRIAL: NCT04538703
Title: Social Media Use of Acne Vulgaris Patients: Multicenter, Survey Work
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Melek Aslan Kayıran, M.D., Istanbul Medeniyet University
Other Study IDs: IstanbulMU7
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: acne vulgaris — Social media use of acne vulgaris patients, a questionnaire will be asked the patients and try to learn how they use social media for getting information about their disease.

SUMMARY:
Acne Vulgaris is a chronic skin disease. However, chronic and repetitive due to the quality of life and psychological status of patients can affect. For this reason, patients carry out various research on their diseases on social media and follow programs on these issues in other media such as television and radio. However, there is no study on how much patients are interested in these publications, how much they trust them, and how they reach and organize information via social media. The aim of the study will be to clarify how and how patients with Acne Vulgaris use social media to obtain information about the diagnosis and treatment of their disease, the interaction of patient groups with each other, and how often social media is used, especially in which group of patients.

ELIGIBILITY:
Inclusion Criteria:

* acne vulgaris patient

Exclusion Criteria:

* who does not want to answer the questions

Ages: 12 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: acne vulgaris patients between 12-60 years of age
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Social media use of acne vulgaris patients, a questionnaire will be asked the patients and try to learn how they use social media for getting information about their disease. | september 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Melek Aslan Kayıran, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided